CLINICAL TRIAL: NCT04240340
Title: Understanding Perceived Barriers to the Disclosure of Psychological Difficulties by Young People With Coeliac Disease
Brief Title: Experiences of Disclosure in Adolescents With Coeliac Disease
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID:14574
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-03

CONDITIONS: Celiac Disease in Children; Celiac Disease; Celiac; Disclosure; Stigma, Social; Emotional Problem; Mental Health Wellness 1
Keywords: coeliac disease; celiac disease; adolescent; wellbeing; mental health; disclosure; stigma
MeSH Terms: conditions — Celiac Disease; Social Stigma; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-structured interview — Semi-structured, face-to-face interviews will be carried out with participants.

SUMMARY:
Being diagnosed with coeliac disease means that individuals can no longer consume things containing gluten, such as bread or cake, or they can become very ill. This can make situations involving food challenging, such as social situations or lunch at school. The investigators know that being diagnosed with coeliac disease as a teenager can be particularly upsetting and can lead to problems such as anxiety or low mood. Research suggests that when young people are worried about the impact of their condition on their life, they can find it challenging to tell their doctor or ask for support.

The investigators would like to understand the experiences of young people with coeliac disease who attend the Paediatric Gastroenterology service at a local children's hospital. The investigators are particularly interested in the reasons why young people either feel able or unable to tell their doctor that they are experiencing difficulties relating to their wellbeing during their appointments, in order to improve support for young people.

This study aims to recruit young people between the ages of 11 and 16, who are attending secondary school, to ask them about the things that make it easier or more difficult to share any concerns about their wellbeing with their doctor.

DETAILED DESCRIPTION:
Background -

Coeliac Disease is a genetic lifelong autoimmune condition whereby ingesting gluten leads to a range of idiosyncratic symptoms including diarrhoea, abdominal pain and chronic fatigue. Treatment for coeliac disease requires the individual to maintain a strict gluten free diet (GFD), whereby the individual must exclude foods containing wheat, barley and rye such as bread, pasta and baked goods.

Research indicates that being diagnosed with coeliac disease as a young person, of secondary school age, poses particular challenges when adapting to the new diet and lifestyle. Developmentally, this age-range involves increasing autonomy from parents, growing responsibility for one's own wellbeing and food related activities and increasing peer-pressure to conform. Consequently, young people with coeliac disease can often experience both felt stigma (the fear of discrimination) and enacted stigma (the experience of discrimination) from their peers. Difficulties adapting to a diagnosis of coeliac disease at this age can lead to non-adherence, poor health related quality of life and psychological difficulties. Indeed, higher rates of anxiety, depression and somatic complaints have been found in young people with coeliac disease, emphasising the importance of early detection of psychological difficulties associated with the condition by services.

This poses as a challenge to services, as young people may also experience increased difficulties disclosing psychological difficulties, which may be exacerbated by the process of adjusting to a chronic condition. For instance, research exploring disclosure and support-seeking in young people with Inflammatory Bowel Disease suggests that, despite a high prevalence of anxiety related to health treatments and psychosocial factors, only half of individuals shared these concerns during routine consultations. A recent systematic review suggests that the characteristics of the potential provider of help, such as credibility, unhelpful responses, being perceived as 'too busy', being perceived as an 'inappropriate source of help for mental distress', unfamiliarity and felt stigma from the source of help itself are possible perceived barriers to help-seeking in 11-25 year olds.

Rationale for the current project -

The recruiting service diagnoses approximately 30 young people with coeliac disease each year and follow-up an additional 75 young people living with the condition. However, only 5 referrals for young people with coeliac disease were made by the Gastroenterology team to Children's Psychological Medicine in 2018.

This raises the question of whether young people with coeliac disease feel that they have had the opportunity to disclose psychological distress associated with coeliac disease during routine consultations, or whether they too perceived barriers to disclosure. This project aims to address these issues systematically by providing a theoretically integrative account of young people's experiences of seeking psychological support from clinicians in the service.

This research project thus has two principal research objectives:

1. To understand perceived barriers to the disclosure of psychological difficulties by young people, aged 11-16 years, with coeliac disease.
2. To make recommendations to the Paediatric Gastroenterology service based on these findings in order to promote disclosure, if it is felt to be helpful, and improve the identification of young people with coeliac disease who may want and benefit from psychological support.

The principal research questions are as follows:

1. What are young people's experiences of disclosing and not disclosing psychological difficulties associated with coeliac disease to clinicians in the service?
2. Could specific changes be made to the service to promote disclosure and improve access to psychological services, if it is felt that this would be helpful for this population?

Broadly, the results of this project could either suggest that young people feel that they had the opportunity to disclose psychological difficulties associated with their condition if they wanted to, or that they did not due to perceived barriers. The latter finding could prompt service improvements from each group in the following ways:

* The service is motivated to implement changes that further integrated care by acknowledging the interdependence among one's biological, social and psychological needs, in line with the 10-year plan. They recognise that the long-term impact of this could reduce non-adherence to the GFD, reduce avoidable medical utilisation and further complications, either medically or with regards to deteriorating mental health.
* Findings could improve young people's experience of the service and access to psychological support. It may also normalise the difficult experience of disclosing distress, affording therapeutic benefit.
* More broadly, this research has the potential to inform NICE guidance around post-diagnosis support for young people with this condition.

Participants:

Participants will be aged between 11 - 16 years and attending secondary school, with a diagnosis of coeliac disease. This age range was selected based on research which suggests that adolescents with coeliac disease are particularly at risk of developing psychological difficulties in relation to their health condition, and can find it particularly difficult to disclose psychological difficulties to healthcare professionals. This is balanced against a need for homogeneity in using IPA. This age range is compatible with the ages of service users presenting in the recruiting service.

Participants recruited will be presenting to the Paediatric Gastroenterology department at a local Children's Hospital, as this project primarily aims to make improvements to this particular service based on its findings. The participants will have received the diagnosis of coeliac disease a minimum of three months prior to participation in the study. This is to allow time for them to process the diagnosis and for treatment to be established. They will also have had at least 1 follow-up appointment following diagnosis, as this will give them an experience to reflect on during the interview. Participants will need to speak fluent English as there is no funding available for interpreters or translation of documents and questionnaires.

Methods:

The chosen methodology for this qualitative study is Interpretive Phenomenological Analysis (IPA). IPA seeks to understand and 'give voice' to the concerns of participants then contextualize and 'make sense' of their worldview from a psychological perspective. IPA has been chosen to meet the studies aims and objectives as it allows the researchers to carry out an in-depth inquiry into the participants' perspectives of possible barriers to disclosing psychological difficulties, with special consideration of the interpersonal and socio-developmental context.

Semi-structured, face-to-face interviews will be carried out, as this is the most appropriate method of data collection for IPA.

Analysis:

Interpretive Phenomenological Analysis will be used as this study seeks to provide an in-depth exploration of the lived experience of individuals with coeliac disease. This will allow researchers to maintain a rich idiographic account of each individual whilst allowing convergence and divergence of themes across transcripts. NVivo may be used to store and organise data, however no software will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Male or Female, aged 11 - 16 years
* Have a medical diagnosis of Coeliac Disease
* Attending Secondary school
* Able to speak fluent English
* Have been under the care of the Paediatric Gastroenterology service at the local Children's Hospital for >3 months and have had >1 follow-up appointment

For participants aged 11-15 only:

* Willing and able to give assent for participation in the study
* Parent/guardian is willing and able to give informed consent for their child's participation in the study

For participants aged 16:

• Willing and able to give consent for participation in the study

Exclusion Criteria:

* Young people with comorbid gastro-intestinal conditions
* Young people currently receiving psychological support from any psychological service.

Ages: 11 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Participants recruited will be presenting to the Paediatric Gastroenterology department at a local Children's Hospital, as this project primarily aims to make improvements to this particular service based on its findings. The participants will have received the diagnosis of coeliac disease a minimum of three months prior to participation in the study. This is to allow time for them to process the diagnosis and for treatment to be established. They will also have had at least 1 follow-up appointment following diagnosis, as this will give them an experience to reflect on during the interview. Participants will need to speak fluent English as there is no funding available for interpreters or translation of documents and questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Semi-structured interview | Lasts up to 90 minutes per participant.
  Includes questions around experiences of having coeliac disease and experiences of disclosing psychological difficulties to clinicians in the service.

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Wheeler, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals Nhs Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be kept for 5 years, separately to any identifiable information, and will then be disposed of securely. This is in accordance with Trust policy. The interviews will be deleted when the research study is finished.

REFERENCES:
- [Background] Ashton, K., Myers, S., Whitehead, E., & Sebastian, S. (2016). OC-058 Perspectives of Adolescent IBD Patients Undergoing Surgery. Gut, 65, A34. doi: 10.1136/gutjnl-2016-312388.57
- [Background] Barratt SM, Leeds JS, Sanders DS. Factors influencing the type, timing and severity of symptomatic responses to dietary gluten in patients with biopsy-proven coeliac disease. J Gastrointestin Liver Dis. 2013 Dec;22(4):391-6. PMID 24369320
- [Background] Green PH, Jabri B. Coeliac disease. Lancet. 2003 Aug 2;362(9381):383-91. doi: 10.1016/S0140-6736(03)14027-5. PMID 12907013
- [Background] Green PH, Jabri B. Celiac disease. Annu Rev Med. 2006;57:207-21. doi: 10.1146/annurev.med.57.051804.122404. PMID 16409146
- [Background] Gulliver A, Griffiths KM, Christensen H. Perceived barriers and facilitators to mental health help-seeking in young people: a systematic review. BMC Psychiatry. 2010 Dec 30;10:113. doi: 10.1186/1471-244X-10-113. PMID 21192795
- [Background] Ludvigsson JF, Agreus L, Ciacci C, Crowe SE, Geller MG, Green PH, Hill I, Hungin AP, Koletzko S, Koltai T, Lundin KE, Mearin ML, Murray JA, Reilly N, Walker MM, Sanders DS, Shamir R, Troncone R, Husby S. Transition from childhood to adulthood in coeliac disease: the Prague consensus report. Gut. 2016 Aug;65(8):1242-51. doi: 10.1136/gutjnl-2016-311574. Epub 2016 Apr 18. PMID 27196596
- [Background] Mayer M, Greco L, Troncone R, Auricchio S, Marsh MN. Compliance of adolescents with coeliac disease with a gluten free diet. Gut. 1991 Aug;32(8):881-5. doi: 10.1136/gut.32.8.881. PMID 1885070
- [Background] Mazzone L, Reale L, Spina M, Guarnera M, Lionetti E, Martorana S, Mazzone D. Compliant gluten-free children with celiac disease: an evaluation of psychological distress. BMC Pediatr. 2011 May 27;11:46. doi: 10.1186/1471-2431-11-46. PMID 21619651
- [Background] NHS England (2019) The NHS Long Term Plan. Retrieved from https://www.longtermplan.nhs.uk/wpcontent/uploads/2019/01/nhs-lo ng-term-plan.pdf
- [Background] NICE. (2015). Clinical Guidelines: Coeliac Disease Recognition, assessment and management: Methods, evidence and recommendations (Standard No. NG20). Retrieved from https://www.nice.org.uk/guidance/ng20/evidence/Full guidance-pdf- 438530077
- [Background] Olsson C, Lyon P, Hornell A, Ivarsson A, Sydner YM. Food that makes you different: the stigma experienced by adolescents with celiac disease. Qual Health Res. 2009 Jul;19(7):976-84. doi: 10.1177/1049732309338722. PMID 19556403
- [Background] Rickwood DJ, Deane FP, Wilson CJ. When and how do young people seek professional help for mental health problems? Med J Aust. 2007 Oct 1;187(S7):S35-9. doi: 10.5694/j.1326-5377.2007.tb01334.x. PMID 17908023
- [Background] Rutter, M., & Smith, D.J. (1995). Psychosocial Disorders in Young People: Time Trends and Their Causes. Chicester: John Wiley & Lons Ltd.
- [Background] Schroeder, R. D., & Mowen, T. J. (2014). "You Can't Eat WHAT?" Managing the Stigma of Celiac Disease. Deviant Behavior, 35(6), 456-474. doi: 10.1080/01639625.2014.855105
- [Background] Smith, J. A., Flowers, P., & Larkin, M. (2009). Interpretative phenomenological analysis: Theory, method and research. London: Sage.